CLINICAL TRIAL: NCT06852742
Title: A Randomized, Evaluator-Blind, Twelve-Week Usage Study to Evaluate and Compare the Efficacy of Two Facial Creams on Moderately to Severely Photodamaged Skin
Brief Title: A Study to Evaluate and Compare the Efficacy of Two Facial Creams on Moderately to Severely Photodamaged Skin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Consumer Inc. (J&JCI) (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: CS2024SK100190
Record Dates: First submitted 2025-01-28; First posted 2025-02-28 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Photodamaged Skin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Facial Cream A (Cell A) (Experimental): Each subject will be provided with the assigned IP (Facial Cream A) and the APs to use for 12 weeks.
  Interventions: Other: Facial Cream A
- Arm 2: Facial Cream B (Cell B) (Experimental): Each subject will be provided with the assigned IP (Facial Cream B) and the APs to use for 12 weeks.
  Interventions: Other: Facial Cream B

INTERVENTIONS:
Other: Facial Cream A — The participants will use the Facial Cleanser twice daily (morning and evening). The Facial Cream A will be applied topically evenly over the entire face after cleansing and drying face in the morning and in the evening. The Sunscreen will be applied evenly over the entire face after Facial Cream A in the morning and re-applied after 80 minutes of swimming or sweating, immediately after towel drying, and at least every 2 hours during sun exposure.
  Arms: Arm 1: Facial Cream A (Cell A)
Other: Facial Cream B — The participants will use the Facial Cleanser twice daily (morning and evening).The Sunscreen will be applied evenly over the entire face after cleansing in the morning and re-applied after 80 minutes of swimming or sweating, immediately after towel drying, and at least every 2 hours during sun exposure. The Facial Cream B will be applied in the evening after washing and drying face.
  Arms: Arm 2: Facial Cream B (Cell B)

SUMMARY:
The objective of this study is to evaluate the efficacy of a retinol alternative-containing facial cream in improving skin texture, radiance/brightness, and the appearance of fine lines, wrinkles, uneven skin tone, and dark spots, with a positive control of a retinol-containing cream.

ELIGIBILITY:
Inclusion Criteria:

* Fitzpatrick Skin Type I, II, III, or IV
* Final review of eligibility (Visit 2): Exhibits moderate to severe (score of 4-7 on a 0-9-point scale) overall photodamage on her face, as evaluated by the PI at Visit 2
* Final review of eligibility (Visit 2): Has a score of at least 4-7 (moderate to severe, on a 0-9-point scale) on at least 3 of the 5 following clinical grading parameters on her face, as evaluated by the PI at Visit 2:

  i. Global fine lines ii. Wrinkles (under-eye and/or crow's feet) iii. Tactile surface roughness iv. Overall unevenness of skin tone v. Lack of radiance/brightness vi. Lack of skin firmness (look and/or feel)
* Generally in good health
* Able to read, write, speak, and understand English
* Individual has signed the Consent for Photograph Release and ICD including Health Insurance Portability and Accountability Act disclosure
* Intends to complete the study and is willing and able to follow all study instructions

Exclusion Criteria:

* Has known allergies or adverse reactions to common topical skincare products or ingredients in the investigational study materials
* Has a pre-existing or dormant facial dermatologic condition that, in the PI or designee's opinion, may confound the study results or otherwise be inappropriate for study participation (e.g., severe acne, acne conglobata, psoriasis, rosacea, rashes, eczema, atopic dermatitis, skin cancer, many and/or severe excoriations, observable suntan/sunburn, scars, nevi, tattoo, excessive hair, etc.)
* Has self-perceived very sensitive skin
* Has self-reported Type 1 or Type 2 diabetes or is taking insulin or another anti-diabetic medication.
* Is taking a medication/using a product that would mask an Adverse Event or confound the study results
* Is self-reported to be pregnant, lactating, or planning to become pregnant during the study or within 30 days of study completion
* Has a history of or a concurrent health/other condition/situation which, in the opinion of the PI, may put the individual at significant risk, confound the study results, or interfere significantly with the individual's participation in the study
* Has a surgery and/or invasive medical procedure planned during the study
* Is simultaneously participating in any other study or has participated in any study within 30 days prior to Visit 1
* Is an employee/contractor or immediate family member of the PI, Study Site, or Sponsor

Ages: 35 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2025-01-20 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Clinical Efficacy Assessment | Visit 5 (Day 84 ± 3)
  Change from baseline on global fine lines, under-eye wrinkles, and crow's feet wrinkles by clinical evaluation. The Principal Investigator will assess each subject's facial condition for the appearance of the mentioned signs on a scale of 0-9, where 0=none, 1-3=mild, 4-6=moderate and 7-9=severe.
Cutaneous Tolerance Assessment | Visit 3 (Day 28 ± 3)
  Change from baseline on erythema, dryness/scaling, burning/stinging, and feeling of dryness/tightness. The Principal Investigator will assess each subject's facial condition for the appearance of the mentioned signs on a scale of 0-3, where 0=none, 1=mild, 2=moderate and 3=severe.

SECONDARY OUTCOMES:
Clinical Efficacy Assessment | Visit 3 (Day 28 ± 3); Visit 4 (Day 56± 3);
  Change from baseline on global fine lines, under-eye wrinkles, and crow's feet wrinkles by clinical evaluation. The Principal Investigator will assess each subject's facial condition for the appearance of the mentioned signs on a scale of 0-9, where 0=none, 1-3=mild, 4-6=moderate and 7-9=severe.
Clinical Efficacy Assessment | Visit 3 (Day 28 ± 3); Visit 4 (Day 56± 3); Visit 5 (Day 84 ± 3)
  Change from baseline on Tactile surface roughness; Lack of clarity; Lack of global firmness (look); Lack of global skin firmness (feel); Elasticity (pinch recoil evaluation);Overall unevenness of skin tone (brown tones); Lack of radiance/brightness; Overall photodamage; Mottled hyperpigmentation; Discrete pigmentation; Skin elasticity/resiliency via pinch-recoil measurement. The Principal Investigator will assess each subject's facial condition for the appearance of the mentioned signs on a scale of 0-9, where 0=none, 1-3= mild, 4-6=moderate and 7-9=severe. For Skin elasticity/resiliency, the Principal Investigator will pinch the skin at the test site between the thumb and middle finger, hold the skin in place for approximately two seconds, and then note the time for the skin to return to its original conformation. A decrease in pinch-recoil times indicates an increase in skin elasticity/resiliency.
Cutaneous Tolerance Assessment | Visit 3 (Day 28 ± 3); Visit 4 (Day 56± 3); Visit 5 (Day 84 ± 3)
  Change from baseline on edema and itching. The Principal Investigator will assess each subject's facial condition for the appearance of the mentioned signs on a scale of 0-3, where 0=none, 1=mild, 2=moderate and 3=severe.
Cutaneous Tolerance Assessment | Visit 4 (Day 56± 3); Visit 5 (Day 84 ± 3)
  Change from baseline on erythema, dryness/scaling, burning/stinging, and feeling of dryness/tightness. The Principal Investigator will assess each subject's facial condition for the appearance of the mentioned signs on a scale of 0-3, where 0=none, 1=mild, 2=moderate and 3=severe.
Self-Assessment | Visit 3 (Day 28 ± 3); Visit 4 (Day 56± 3); Visit 5 (Day 84 ± 3)
  Participant's self-assessment questionnaire to assess the facial skin condition. Participants will answer six questions and rate their responses on a scale from 1 to 10, where a higher score indicates a more positive response.
Product Assessment | Visit 3 (Day 28 ± 3); Visit 4 (Day 56± 3); Visit 5(Day 84 ± 3)
  Product assessment questionnaire to assess the percentage of favorable responses compared to unfavorable responses. Participants will answer 23 questions and rate as: Disagree completely, disagree somewhat, neither agree nor disagree, agree somewhat and agree completely.

CONTACTS AND LOCATIONS:
Locations (1):
- KGL Skin Study Center, LLC, West Chester, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No